CLINICAL TRIAL: NCT06926972
Title: NOURISH: NutritiOUs fRuIts and veggieS to Improve Health: A Culinary Medicine Intervention
Brief Title: NutritiOUs fRuIts and veggieS to Improve Health: A Culinary Medicine Intervention
Acronym: NOURISH
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-23506
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cancer, Nos
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NOURISH: NutritiOUs fRuIts and veggieS to improve Health (Experimental): Intervention Phase: In the intervention phase, members of the John Geigle YMCA will be assigned to the NOURISH intervention, which includes biweekly provision of f/v, recipe cards, and nutritional education handouts plus 30-minute culinary medicine demonstrations with skill-building training (six total demonstrations focused on f/v recipes). Members of the Hernando County YMCA will be assigned to the control condition and participants will receive recipe cards and nutritional education handouts but will not receive f/v or cooking demonstrations.
  Maintenance Phase: In the maintenance phase, we will better understand adherence to dietary guidelines once f/v are no longer provided and maintenance of culinary skills.
  Interventions: Other: NOURISH

INTERVENTIONS:
Other: NOURISH — Culinary medicine demonstrations and nutritional education focused on balanced eating.

SUMMARY:
This study includes a 12-week culinary medicine intervention integrated within the existing YMCA Suncoast Survivorship and Wellness Program Powered by Moffitt. Members of the John Geigle YMCA will be assigned to the NOURISH intervention, which includes biweekly provision of fruit and vegetable bundles, recipe cards, and nutritional education handouts plus 30-minute culinary medicine demonstrations with skill-building training (six total demonstrations focused on fruit and vegetable recipes).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer.
* Able to speak and read English.
* Without documented or observable psychiatric or neurologic diagnoses that could interfere with participation (e.g., dementia, active psychosis).
* Able to provide informed consent.

Exclusion Criteria:

* Not meeting all of the above inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Participant Recruitment Rate | Up to 1 year
  Number of participants successfully recruited to the study.
Participant Retention | Up to 1 year
  The proportion of participants who complete the study.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Crowder, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States